CLINICAL TRIAL: NCT00743366
Title: Effect of Quetiapine on Marijuana Withdrawal and Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5685; 5P50DA009236 (NIH)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Marijuana Smoking
Keywords: quetiapine; smoked marijuana; marijuana use
MeSH Terms: conditions — Marijuana Smoking; Marijuana Use | interventions — nabiximols; Quetiapine Fumarate; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine (200mg/day), Marijuana (6.2%, 0.0%) (Experimental): Quetiapine (200mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (200 mg) were administered 2 times per day ((1100 and 2300 hours).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Marijuana; Drug: Quetiapine
- Placebo, Marijuana (6.2%, 0.0%) (Placebo Comparator): Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Marijuana; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Marijuana — 0,6.2% THC
  Other Names: cannabis
Drug: Quetiapine — 200 mg/day
  Other Names: seroquel
  Arms: Quetiapine (200mg/day), Marijuana (6.2%, 0.0%)
Drug: Placebo oral capsule
  Other Names: Riboflavin
  Arms: Placebo, Marijuana (6.2%, 0.0%)

SUMMARY:
The objective of this study is to investigate the interaction between marijuana and quetiapine, with the goal of using this information to improve marijuana treatment outcome.

DETAILED DESCRIPTION:
The purpose of this study is to determine if quetiapine decreases marijuana relapse in a controlled lab setting. For the purposes of this model, relapse is defined as a return to marijuana use after a period of abstinence. The study will utilize an inpatient/outpatient, counter-balanced design, with each participant maintained on placebo and quetiapine (200 mg/day) for 18 days. Participants will begin taking capsules as outpatients so that the dose can be incremented prior to the inpatient phase. While inpatient, participants will have the opportunity to self-administer placebo (0.0%) or active marijuana (6.2%) 6 times per day, depending on the study day. Our laboratory model, which has distinguished the effects of a range of medications on marijuana withdrawal and relapse, will provide important information on the effect of quetiapine as a potential short-term pharmacotherapy to facilitate abstinence in the initial stages of marijuana treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use:average of 2 marijuana cigarettes per day at least 4 times per week for the past 4 weeks
* Able to perform study procedures
* 21-45 years of age
* Women practicing an effective form of birth control (condoms, diaphragm, birth control, pill, IUD)
* Normal body weight

Exclusion Criteria:

* Current, repeated illicit drug use (other than marijuana)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension, clinically significant abnormalities)
* History of heart disease or current conduction system disease as indicated by QRS duration > 0.11
* Request for drug treatment
* Current parole or probation
* Pregnancy or current lactation
* Recent history of significant violent behavior
* Major current Axis I psychopathology (major depressive disorder, bipolar disorder, suicide risk, schizophrenia)
* Current use of any prescription or over-the-counter medication
* Prior allergic or otherwise serious adverse reaction to quetiapine

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Cooper ZD, Foltin RW, Hart CL, Vosburg SK, Comer SD, Haney M. A human laboratory study investigating the effects of quetiapine on marijuana withdrawal and relapse in daily marijuana smokers. Addict Biol. 2013 Nov;18(6):993-1002. doi: 10.1111/j.1369-1600.2012.00461.x. Epub 2012 Jun 28. PMID 22741619

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 volunteers completed the study (12 males; 2 females). An additional 6 volunteers enrolled (5 males, 1 female), but did not complete.
Groups:
- Quetiapine (200mg/Day), Placebo: Quetiapine (200mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (200 mg) were administered 2 times per day (1100 and 2300 hours).
- Placebo, Quetiapine (200mg/Day): Placebo medication (2x/day): Packaged riboflavin in size 00 opaque capsules to match size of active medication. Placebo capsules were administered 2 times per day (1100 and 2300 hours).
Period: Intervention 1 (8 Days)
Arm/Group | Quetiapine (200mg/Day), Placebo | Placebo, Quetiapine (200mg/Day)
Started | 10 | 10
Completed | 7 (A total of 6 participants withdrew before completion of the final inpatient phase) | 7 (A total of 6 participants withdrew before completion of the final inpatient phase)
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3
Period: Intervention 2 (8 Days)
Arm/Group | Quetiapine (200mg/Day), Placebo | Placebo, Quetiapine (200mg/Day)
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Measure of Relapse: Change in Puffs Chosen Between Baseline and Relapse Phase
Description: This is a measure of marijuana self-administration and relapse since each initial puff costs $10 and is a burden to overcome just to smoke.
  Over each 3 day period, the puffs chosen by each participant is averaged for a single value.
Time Frame: Days 1-3 (Baseline) and Days 6-8 (Relapse Phase)
Measure: Mean (Standard Error); unit: Puffs
Groups:
- Quetiapine, Marijuana: quetiapine's effects on marijuana withdrawal and relapse
  Marijuana: 0,6.9% THC
  Quetiapine: 0, 200 mg/day
Arm/Group | Quetiapine, Marijuana | Placebo, Marijuana
Number analyzed (Participants) | 14 | 14
Puffs | 2.5 (0.6) | 1.5 (1.1)

ADVERSE EVENTS:
Arm/Group | Quetiapine (200mg/Day), Placebo | Placebo, Quetiapine (200mg/Day)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (200mg/Day), Placebo (N=20) | Placebo, Quetiapine (200mg/Day) (N=20)
gastrointestinal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) — gastrointestinal discomfort (nausea, vomiting, stomach pain, constipation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No